CLINICAL TRIAL: NCT06653179
Title: Comparison of the Efficacy of Sacral Erector Spinae Plane Block and Caudal Epidural Injection on Chronic Coccydynia: A Randomized Controlled Trial
Brief Title: Efficacy of Interventional Methods Used in the Treatment of Coccydynia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Turan, MD, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sacral ESP vs Caudal Epidural
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Coccydynia; Erector Spinae Plane Block; Caudal Block
Keywords: Sacral Erector Spinae Plane Block; Caudal. Epidural Injection; Chronic Coccydynia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral Erector Spinae Plane Block Group (Active Comparator): Sacral Erector Spinae Plane Block for Chronic Coccydynia
  Interventions: Procedure: Sacral Erector Spinae Plane Block
- Caudal Epidural Injection Gropu (Active Comparator): Caudal Epidural Injection for Chronic Coccydynia
  Interventions: Procedure: Caudal Epidural Injection

INTERVENTIONS:
Procedure: Sacral Erector Spinae Plane Block — The patient is placed in the prone positionon a procedure table. The sacral region is exposed, and the area is prepped with antiseptic solution under sterile conditions. The ultrasound high-frequency linear transducer is placed transversely over the sacrum. The sacral cornua are typically seen as bony structures adjacent to the sacral hiatus, appearing as two hyperechoic structures. Rotate the ultrasound probe to a sagittal position over the sacrum to align with the fourth and fifth sacral vertebrae. Under continuous ultrasound guidance, block needle is inserted in-plane with the ultrasound probe. Direct the needle through the soft tissue towards the plane between the erector spinae muscle and the sacrum. After confirming needle placement, the injectate mixture of 8 mg dexamethasone and 10 mg bupivacaine (0.5% concentration) is administered. A total volume of 10 mL is injected, and real-time ultrasound is used to observe the spread of the injectate within the target tissue plane.
  Arms: Sacral Erector Spinae Plane Block Group
Procedure: Caudal Epidural Injection — The patient is positioned in the prone position on the procedure table, and the sacral region is exposed and prepped with antiseptic solution under sterile conditions. The fluoroscope is positioned laterally to visualize the sacral hiatus. Under fluoroscopic guidance, the block needle is inserted through the skin and advanced toward the sacral hiatus. Continuous fluoroscopy is used to ensure correct needle placement, typically visualized at the level of the sacral canal. After confirming the appropriate position with contrast media, the injectate consisting of 8 mg dexamethasone and 10 mg bupivacaine (0.5% concentration) is slowly administered, with a total volume of 10 mL. During injection, careful monitoring of the needle position is performed to avoid intravascular injection. After the procedure, patients are monitored for potential complications such as hypotension and allergic reactions.
  Arms: Caudal Epidural Injection Gropu

SUMMARY:
This study aims to evaluate the effectiveness of sacral erector spinae plane block and caudal epidural injection in patients with coccydynia resistant to conservative treatments. Ultrasound guidance will be used for sacral erector spinae plane block, while fluoroscopic guidance will be applied for caudal epidural injection. The effectiveness of these treatments will be assessed through face-to-face questionnaires, the Numerical Rating Scale and the Paris Functional Coccydynia Scale at first, fourth and twelfth-week follow-ups.

DETAILED DESCRIPTION:
Coccydynia (coccygodynia, coccalgia) or coccygeal pain is a painful syndrome affecting the coccyx region. The most important etiological factors in the formation of coccydynia are external and internal trauma, though it can also occur idiopathically. The pain intensifies while sitting or standing up from a sitting position. Although it can affect individuals of all ages and genders, the average onset age is 40, with a prevalence 5 times higher in women. Coccydynia is a painful condition that impacts quality of life, and its treatment can be challenging due to the influence of various physiological and psychological factors.

Patients typically complain of pain in the tailbone area, which increases with prolonged sitting, leaning backward while sitting, standing for extended periods, and rising from a sitting position. Conservative treatments such as nonsteroidal anti-inflammatory drugs, levator ani relaxation exercises, seating cushions, and transcutaneous electrical stimulation are commonly used, but these methods are ineffective in 10% of cases.

For patients unresponsive to conservative treatments, interventional and surgical options include caudal epidural steroid injection, sacral erector spinae plane block, ganglion impar blocks, radiofrequency ablation of sacral nerves, block and radiofrequency ablation of coccygeal nerves, and coccygectomy.

Sacral erector spinae plane block under ultrasound guidance or caudal epidural injection under fluoroscopic guidance is performed under sterile conditions for patients with resistant and chronic coccydynia. For the sacral erector spinae plane block, the sacral and coccygeal cornua are visualized in a transverse position under ultrasound, followed by sagittal positioning of the probe over the sacrum for injection at the 4th and 5th sacral vertebrae. For caudal epidural injection, the fluoroscope is positioned laterally, and the injection is administered to the target area under fluoroscopic imaging. In both techniques, the injectate consists of 8 mg dexamethasone and 10 mg bupivacaine (0.5% concentration), with a total volume of 10 mL. After the procedure, patients are monitored for potential hypotension and allergic reactions as a precaution.

This study will include patients treated with sacral erector spinae plane block and caudal epidural injection for coccydynia resistant to conservative treatments. Face-to-face questionnaires, Numerical Rating Scale scores, and the Paris Functional Coccydynia Scale will be evaluated at 1, 4, and 12-week follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coccydynia unresponsive to conservative treatment
* Male and female population aged 18-70
* No previous interventional procedure performed during the treatment process

Exclusion Criteria:

* Coagulation disorders
* Infections in the areas to be treated
* Allergy to local anesthesia
* Socio-cultural inadequacy
* Mental retardation
* Pregnancy
* Previous interventional procedure performed
* Patient refusal of the interventional procedure
* Presence of malignancy in the coccygeal region
* Previous surgery in the coccygeal region

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Change from baseline to 1st and 2nd and twelfth week after treatment
  Numeric Rating Scale is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)
Paris Functional Coccydynia Scale | Change from baseline to 1st and 2nd and twelfth week after treatment
  The Paris Functional Coccydynia Scale is designed to assess the functional impact of coccydynia on patients' daily lives. It comprises various items that evaluate pain intensity, functional limitations, and the effect of pain on daily activities. Scores range from 0 to 10, with higher scores indicating greater impairment and more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Etlik, Turkey (Türkiye)